CLINICAL TRIAL: NCT02932605
Title: Endocannabinoid Control of Microglia Activation as a New Therapeutic Target in the Treatment of Schizophrenia
Acronym: CANGLIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, M.G. Bossong, Assistant Professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ABR58805; 2016-003529-41 (EudraCT Number)
Record Dates: First submitted 2016-09-21; First posted 2016-10-13 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cannabidiol; Magnetic Resonance Spectroscopy (1H-MRS); Microglia
MeSH Terms: conditions — Schizophrenia | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): Patients will be treated with 600mg CBD daily for 4 weeks (28 days)
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Patients will be treated with placebo daily for 4 weeks (28 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Cannabidiol — Cannabidiol
  Arms: Cannabidiol

SUMMARY:
The main objective of this study is to compare microglia activation as measured with proton Magnetic Resonance Spectroscopy (1H-MRS) between recent-onset schizophrenia patients who are randomised to CBD and those randomised to placebo.

DETAILED DESCRIPTION:
Schizophrenia is a chronic and severe mental disorder with an urgent need for new and more effective treatments. A promising novel pharmacological target in this respect is the endocannabinoid system. In particular the cannabinoid compound cannabidiol (CBD) displays a highly favourable profile for development as a new antipsychotic agent. Increasing evidence indicates a significant role for neuroinflammation in the pathophysiology of schizophrenia, especially for activation of resident macrophages of the brain: microglia. Interestingly, converging preclinical evidence suggests that microglia activation is under control of the endocannabinoid system. However, how manipulation of the endocannabinoid system affects microglia activation in humans has not been established, but it is presumably related to clinical improvement of schizophrenia patients.

In this project, we propose to study endocannabinoid control of microglia activation as a new therapeutic target in the treatment of schizophrenia. Using a placebo-controlled, randomised, double-blind design, we will investigate this in a group of 36 recent-onset schizophrenia patients after four weeks of daily CBD treatment, in addition to their regular antipsychotic medication. First, we will examine if CBD treatment attenuates microglia activation and levels of peripheral inflammatory markers. In vivo microglia activation is assessed before and after treatment using 1H-MRS, with the level of myo-inositol being regarded as a marker of glia function. Second, we will determine if reduced microglia activation and levels of inflammatory markers relate to improvement of symptomatology and cognitive function. Third, we will assess how microglia activation and levels of inflammatory markers before treatment predict the clinical response to CBD.

ELIGIBILITY:
Inclusion Criteria:

* A DSM-IV diagnosis of 295.x (schizophrenia, schizophreniform disorder or schizoaffective disorder) or 298.9 (psychosis NOS). Diagnosis must be confirmed in writing by the treating psychiatrist.
* Age 16 - 40
* Onset of first psychosis no longer than five years ago
* Written informed consent of the subject

Exclusion Criteria:

* Any clinically significant medical condition that may influence the results of the trial or affect the ability to take part in a trial
* Routine laboratory screening values considered an impediment for participation by a medical doctor (see Appendix 1)
* Positive urine test on any drug of abuse, except cannabis
* Treatment with more than one antipsychotic agent or with an unstable dose of one type of antipsychotic medication in the month prior to study inclusion
* Use of glucocorticosteroids or non-steroidal anti-inflammatory drugs (NSAIDs) within two weeks prior to study inclusion
* Use of co-medication other than antipsychotics that has a clinically relevant interaction with the cytochrome P450 (CYP) 2C19 or CYP3A classes of liver enzymes within two weeks prior to study inclusion (because CBD may be an inhibitor of these classes of liver enzymes; see paragraph 6.3)
* Intake of investigational drug within one month prior to study inclusion
* Daily use of alcohol or drugs of abuse (including cannabis) in the three months prior to study inclusion
* Any current or previous neurological disorder, including epilepsy
* History of head injury resulting in unconsciousness lasting at least 1 hour
* IQ < 70, as measured with Dutch version of the National Adult Reading Test (DART)
* Breastfeeding, pregnancy or attempting to conceive
* MRI contraindications, e.g. claustrophobia or metal objects in or around the body

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
the concentration of prefrontal metabolites as measured with 1H-MRS | 4 weeks
  the concentration of prefrontal metabolites as measured with 1H-MRS, with the level of myo-inositol being regarded as a marker of glia function

SECONDARY OUTCOMES:
Tolerability associated with CBD treatment | 4 weeks
  Number of treatment-related adverse events as assessed by the study physician
Psychotic symptoms | 4 weeks
  Measured with the Positive and Negative Syndrome Scale (PANSS)
Depressive symptoms | 4 weeks
  Measured with the Hamilton Depression Rating Scale (HAM-D)
Anxiety | 4 weeks
  Measured with the State-Trait Anxiety Inventory (STAI)
Clinical impression | 4 weeks
  Measured with the Clinical Global Impressions Scale (CGI)
Psychosocial functioning | 4 weeks
  Measured with the Global Assessment of Functioning scale (GAF)
Social and Occupational functioning | 4 weeks
  Measured with the Social and Occupational Functional Assessment Scale (SOFAS)
Role functioning | 4 weeks
  Measured with the Global Functioning Role (GF:R) scale
Social functioning | 4 weeks
  Measured with the Global Functioning Social (GF:S) scale
Cognitive function | 4 weeks
  Measured with the Brief Assessment of Cognition in Schizophrenia (BACS)
CBD plasma concentrations | 4 weeks
Blood cytokine concentrations | 4 weeks
  Examples of cytokines that could be assessed in the current study include but are not restricted to interferon-γ, interleukin (IL)-1α, IL-1RA, IL-6, IL-10, IL-12, IL-15, tumour necrosis factor-α, and S100B
Haematological blood parameters | 4 weeks
  Platelet activation and platelet aggregate formation are measured
MRI measures | 4 weeks
  Brain structure and function

CONTACTS AND LOCATIONS:
Overall Officials: Matthijs Bossong, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No